CLINICAL TRIAL: NCT04329806
Title: Sympathetic Mechanisms in the Cardiovascular and Metabolic Alterations of Obesity
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study being replaced by crossover design
Sponsor: Italo Biaggioni (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Italo Biaggioni, Professor, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 190479; R01HL149386 (NIH)
Record Dates: First submitted 2020-03-16; First posted 2020-04-01 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Obesity-Associated Insulin Resistance
MeSH Terms: interventions — moxonidine; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moxonidine (Experimental): Moxonidine to be administered at a dose to produce a decrease in BP of at least 20% of baseline for 9 weeks
  Interventions: Drug: Moxonidine 0.2 MG
- Amlodipine (Active Comparator): Amlodipine to be administered at a dose to produce a decrease in BP of at least 20% of baseline for 9 weeks
  Interventions: Drug: Amlodipine 5 MG

INTERVENTIONS:
Drug: Moxonidine 0.2 MG — Moxonidine 0.2 MG twice daily
  Arms: Moxonidine
Drug: Amlodipine 5 MG — Amlodipine 5 MG twice daily
  Arms: Amlodipine

SUMMARY:
The purpose of this study is to study the role of sympathetic mechanisms involved in chronic regulation of cardiovascular and metabolic abnormalities seen in obesity. The investigators will study the effects chronic sympathetic inhibition on insulin sensitivity, inflammation and endothelial function in obese hypertensive human subjects.

DETAILED DESCRIPTION:
Continuing Review (CR, 2021/08/04) Update: Removal of the angiotensin receptor blockade arm of the study

The presence of obesity increases the risk for hypertension and diabetes, in part due to the development of insulin resistance. Obesity is also associated with sympathetic activation and the overarching hypothesis is that sympathetic activation contributes to insulin resistance with impairment of its vascular and metabolic actions. Preliminary studies suggest that 1) Blood pressure can be normalized by autonomic blockade in obese hypertensives, 2) Sympathetic activation provides no metabolic benefit because the increase in resting energy expenditure associated with obesity is due to an increase in fat free mass rather than sympathetic activation. On the contrary, autonomic blockade: 3) Improves insulin sensitivity in obese hypertensives, 4) Reverses their impaired NO-mediated dilation, and 5) Reduces plasma isoprostanes, a measure of oxidative stress. Furthermore, these abnormalities are interrelated in negative feedback loops, whereby inflammation/oxidative stress impairs nitric oxide mechanisms, which in turn reduces insulin-mediated vasodilation important for substrate delivery, thus contributing to insulin resistance; insulin resistance leads to compensatory increases in insulin levels, which contributes to further sympathetic activation. Current treatment guidelines do not specifically address the treatment of obesity hypertension, and do not target sympathetic activation as a first line approach. It is important, therefore, to determine whether or not targeting sympathetic activation offers unique advantages in the treatment of obesity hypertension over current approaches. The investigators propose a proof-of-concept mechanistic study comparing the metabolic, vascular, and anti-inflammatory effects of sympathetic inhibition, calcium channel blockade and angiotensin receptor blockade in obesity hypertension. The investigators will test the hypotheses that sympathetic activation contributes to 1) metabolic insulin resistance, which impairs the suppression of endogenous glucose production and the stimulation of glucose uptake normally provided by insulin, 2) vascular insulin resistance, which impairs insulin-mediated vasodilation and microvascular recruitment that normally promote glucose uptake, and 3) inflammation and oxidative stress, which contribute to insulin resistance and hypertension. The proposed studies will gauge the contribution of sympathetic activation to the cardiovascular and metabolic complications of obesity and provide the mechanistic insight to determine whether or not it should foster the efforts currently under way to develop novel therapies targeting sympathetic activation for hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races between 18 and 60 years of age
* Hypertension defined by two or more properly measured seated blood pressure readings >130/85 mmHg or currently on antihypertensive medication.
* Obesity will be defined as having a body mass index (BMI) ≥ 30 kg/m2.
* Able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy or breast feeding
* Current smokers or history of heavy smoking (>2 packs/day)
* History of alcohol or drug abuse
* Previous allergic reaction to study medications
* Evidence of type I diabetes
* Cardiovascular disease other than hypertension
* History of serious cerebrovascular disease
* History or presence of immunological or hematological disorders
* Impaired renal function
* Treatment with any investigational drug in the 1 month preceding the study
* Inability to give, or withdraw, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moxonidine | Amlodipine
Started | 5 | 5
Completed | 2 | 1
Not Completed | 3 | 4
Not completed — Physician Decision | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxonidine | Amlodipine | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (5) | 41 (6) | 42 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: Dose response curve to insulin (measure as glucose infusion rate, mg/kg/min)
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: mg/kg/min
Groups:
- Moxonidine: Moxonidine to be administered at a dose to produce a decrease in BP of at least 20% of baseline for 9 weeks
  Moxonidine 0.2 MG: Moxonidine 0.2 MG twice daily
  The main outcome is insulin sensitivity (measured as glucose infusion rate in mg/kg/min during the last 30 minutes of the clamp).
- Amlodipine: Amlodipine to be administered at a dose to produce a decrease in BP of at least 20% of baseline for 9 weeks
  Amlodipine 5 MG: Amlodipine 5 MG twice daily
  The main outcome is insulin sensitivity (measured as glucose infusion rate in mg/kg/min during the last 30 minutes of the clamp).
Arm/Group | Moxonidine | Amlodipine
Number analyzed (Participants) | 4 | 4
mg/kg/min | 4.3 (3.1) | 3.6 (3.3)

ADVERSE EVENTS:
Time Frame: For the duration of the study (3 months).
Arm/Group | Moxonidine | Amlodipine
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT04329806/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT04329806/ICF_001.pdf